CLINICAL TRIAL: NCT00670566
Title: Irbesartan/Hydrochlorothiazide to Control Elevated Blood Pressure to Target in Moderate to Severe Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRBEH_L_03170
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: irbesartan/hydrochlorothiazide

INTERVENTIONS:
Drug: irbesartan/hydrochlorothiazide — 50/12.5mg for 4 weeks follow 300/12.5mg for 4 weeks and proceed to 300/25mg for 4 weeks
  Other Names: CoAprovel

SUMMARY:
The primary objective is to evaluate the antihypertensive efficacy of a fixed combination of Irbesartan/HydroChloroThiazide (CoAprovel) in Chinese moderate to severe hypertensive patients.

The secondary objective is to get systolic blood pressure and diastolic blood pressure goal attainment rate from CoAprovel in Chinese hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertensive patients
* Moderate to severe Patients with uncontrolled blood pressure (systolic blood pressure ≥160mmHg, diastolic blood pressure ≥100mmHg for untreated, systolic blood pressure ≥150mmHg, diastolic blood pressure ≥95mmHg for treated on monotherapy).
* Patients are willing to discontinue previous antihypertensive medicine

Exclusion Criteria:

* Pregnant or lactating women, or women of child bearing potential without contraceptive method.
* Hypersensitivity to any component of the products or other sulfonamide derived substances.
* Secondary hypertension.
* Severe renal impairment (Creatinine Clearance ≤30ml/min)
* Severe hepatic impairment, biliary cirrhosis and cholestasis.
* Refractory hypokalemia, hypercalcaemia.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with controlled blood pressure | At month 3

SECONDARY OUTCOMES:
Adverse events | Throughout the study period
Systolic and Diastolic Blood Pressure | At month 3 versus baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mei Mao, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Shanghai, China

REFERENCES:
- [Derived] Ye XF, Wang WY, Wang XY, Huang QF, Li Y, Wang JG. Alcohol Consumption and Antihypertensive Treatment Effect in Male Patients With Hypertension. Am J Hypertens. 2024 Jan 16;37(2):112-119. doi: 10.1093/ajh/hpad091. PMID 37769181